CLINICAL TRIAL: NCT06980090
Title: Neural Mechanisms of Interpersonal Expectations on Negative Affect
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Trustees of Dartmouth College (Other)
Responsible Party: Principal Investigator, Tor Wager, Diana L. Taylor Distinguished Professor, Trustees of Dartmouth College
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 467251
Record Dates: First submitted 2025-05-09; First posted 2025-05-20 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Negative Affectivity; Non-invasive Brain Stimulation; Placebo Effect; Expectations
Keywords: Transcranial temporal interference stimulation; Pain; Fear; Cognitive effort
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: Experiment 1 involves participants completing all conditions formed by combinations of active vs. sham transcranial temporal interference stimulation (tTIS) and positive vs. negative placebo manipulations. The order of sessions is counterbalanced using a Balanced Latin Square approach to minimize order effects, with each participant serving as their own control.
  Experiment 2 specifically focuses on placebo manipulation effects. Participants complete two experimental sessions-one with placebo intervention (On-Placebo) and one without (Off-Placebo)-both sessions utilizing sham tTIS. Session order is counterbalanced, enabling each participant to act as their own control to isolate and assess the effects of the placebo manipulation.
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Experiment 1 - Crossover Order: Session A-B-C-D (Experimental): Participants complete all four experimental sessions in the following sequence: 1. Session A; 2. Session B; 3. Session C; 4.Session D
  Interventions: Behavioral: Session A: Positive Placebo + Active tTIS; Behavioral: Session B: Positive Placebo + Sham tTIS; Behavioral: Session C: Negative Placebo + Active tTIS; Behavioral: Session D: Negative Placebo + Sham tTIS
- Experiment 1- Crossover Order: Session B-C-D-A (Experimental): Participants complete all four experimental sessions in the following sequence: 1. Session B; 2. Session C; 3. Session D; 4. Session A
  Interventions: Behavioral: Session A: Positive Placebo + Active tTIS; Behavioral: Session B: Positive Placebo + Sham tTIS; Behavioral: Session C: Negative Placebo + Active tTIS; Behavioral: Session D: Negative Placebo + Sham tTIS
- Experiment 1- Crossover Order: Session C-D-A-B (Experimental): Participants complete all four experimental sessions in the following sequence: 1. Session C; 2.Session D; 3. Session A; 4. Session B
  Interventions: Behavioral: Session A: Positive Placebo + Active tTIS; Behavioral: Session B: Positive Placebo + Sham tTIS; Behavioral: Session C: Negative Placebo + Active tTIS; Behavioral: Session D: Negative Placebo + Sham tTIS
- Experiment 1- Crossover Order: Session D-A-B-C (Experimental): Participants complete all four experimental sessions in the following sequence: 1. Session D; 2. Session A; 3. Session B; 4. Session C
  Interventions: Behavioral: Session A: Positive Placebo + Active tTIS; Behavioral: Session B: Positive Placebo + Sham tTIS; Behavioral: Session C: Negative Placebo + Active tTIS; Behavioral: Session D: Negative Placebo + Sham tTIS
- Experiment 2 - Crossover Order : Session E-F (Experimental): Participants complete all two experimental sessions in the following sequence: 1. Session E; 2. Session F
  Interventions: Behavioral: Session E: On-Placebo + Sham tTIS; Behavioral: Session F: Off-Placebo + Sham tTIS
- Experiment 2 - Crossover Order : Session F-E (Experimental): Participants complete all two experimental sessions in the following sequence: 1. Session F; 2. Session E
  Interventions: Behavioral: Session E: On-Placebo + Sham tTIS; Behavioral: Session F: Off-Placebo + Sham tTIS

INTERVENTIONS:
Behavioral: Session A: Positive Placebo + Active tTIS — Participants receive active tTIS, with two signals set at 2000 Hz and 2080 Hz, creating an 80 Hz interference beat targeting the anterior/mid-cingulate cortex (aMCC). Stimulation is delivered at 2 mA for 20 minutes. The stimulation is combined with a positive social placebo intervention delivered by the care provider. Participants complete three multimodal negative affect tasks (MNAT) before and after the stimulation.
  Arms: Experiment 1 - Crossover Order: Session A-B-C-D; Experiment 1- Crossover Order: Session B-C-D-A; Experiment 1- Crossover Order: Session C-D-A-B; Experiment 1- Crossover Order: Session D-A-B-C
Behavioral: Session B: Positive Placebo + Sham tTIS — Participants receive sham tTIS, using two identical 2000 Hz signals that produce no low-frequency interference. The device mimics active parameters (2 mA, 20 minutes) without delivering effective stimulation. The sham stimulation is paired with a positive social placebo intervention. Participants complete three MNAT tasks before and after the session.
  Arms: Experiment 1 - Crossover Order: Session A-B-C-D; Experiment 1- Crossover Order: Session B-C-D-A; Experiment 1- Crossover Order: Session C-D-A-B; Experiment 1- Crossover Order: Session D-A-B-C
Behavioral: Session C: Negative Placebo + Active tTIS — Participants receive active tTIS (2000 Hz and 2080 Hz signals, 2 mA, 20 minutes) combined with a negative social placebo intervention (neutral or skeptical messaging about treatment efficacy). Participants complete three MNAT tasks before and after the stimulation.
  Arms: Experiment 1 - Crossover Order: Session A-B-C-D; Experiment 1- Crossover Order: Session B-C-D-A; Experiment 1- Crossover Order: Session C-D-A-B; Experiment 1- Crossover Order: Session D-A-B-C
Behavioral: Session D: Negative Placebo + Sham tTIS — Participants receive sham tTIS (identical 2000 Hz signals, mimicking active stimulation) combined with a negative social placebo intervention. Participants complete three MNAT tasks before and after the session.
  Arms: Experiment 1 - Crossover Order: Session A-B-C-D; Experiment 1- Crossover Order: Session B-C-D-A; Experiment 1- Crossover Order: Session C-D-A-B; Experiment 1- Crossover Order: Session D-A-B-C
Behavioral: Session E: On-Placebo + Sham tTIS — Participants receive sham tTIS (brief 15-second stimulation followed by no current) paired with a positive social placebo intervention. Participants complete three MNAT tasks before and after the session.
  Arms: Experiment 2 - Crossover Order : Session E-F; Experiment 2 - Crossover Order : Session F-E
Behavioral: Session F: Off-Placebo + Sham tTIS — Participants receive sham tTIS (brief 15-second stimulation, then no current) without any placebo intervention. Participants complete three MNAT tasks before and after the session.
  Arms: Experiment 2 - Crossover Order : Session E-F; Experiment 2 - Crossover Order : Session F-E

SUMMARY:
The goal of this clinical trial is to learn whether non-invasive brain stimulation, called transcranial temporal interference stimulation (tTIS), can reduce negative affect, and how expectations shaped by care providers influence these effects.

The main questions this study aims to answer are: (1)Does active tTIS reduce negative affect more effectively than sham (inactive) tTIS? (2)Do positive treatment expectations enhance the effects compared to negative expectations?

Participants will: (1) Receive either active or sham tTIS. (2) Be provided with positive or negative messaging regarding treatment effectiveness. (3) Interact with care providers and complete assessments measuring negative affect and physiological responses.

DETAILED DESCRIPTION:
The study employs a within-subject, crossover factorial design, consisting of two experiments.

Experiment 1

In Experiment 1, 30 participants ('patients') will complete all combinations of two independent variables-stimulation type (active vs. sham tTIS) and placebo manipulation (positive vs. negative placebo messaging)-resulting in four sessions:

* Session A: Positive Placebo + Active tTIS
* Session B: Positive Placebo + Sham tTIS
* Session C: Negative Placebo + Active tTIS
* Session D: Negative Placebo + Sham tTIS

Participants complete three multimodal negative affect tasks (MNAT) before and after each stimulation session. Active tTIS delivers two signals at 2000 Hz and 2080 Hz, generating an 80 Hz interference beat targeted at the anterior/mid-cingulate cortex (aMCC) at 2 mA for 20 minutes. Sham tTIS uses identical frequencies (2000 Hz and 2000 Hz) with no effective interference.

Sessions are administered in a counterbalanced order based on a Balanced Latin Square to minimize order effects, with at least 48 hours between sessions. Participants thus serve as their own controls.

Experiment 2

Experiment 2 includes 160 participants divided into two groups: 120 'patients' and 40 'doctors'.

A within-subject crossover design is employed, focusing specifically on placebo manipulation effects. Patients complete two experimental sessions involving sham tTIS only:

* Session E: On-Placebo + Sham tTIS (with social placebo intervention)
* Session F: Off-Placebo + Sham tTIS (without placebo intervention)

In both sessions, patients complete the same MNAT tasks before and after stimulation. Sham tTIS involves a brief 15-second stimulation followed by no current for the remainder of the session, preserving the illusion of active stimulation.

'Doctors' are trained to administer the sham stimulation and deliver the placebo manipulation. During placebo induction sessions, providers simulate a "personalization" procedure, adjusting sham parameters while covertly reducing pain stimulus intensity to enhance placebo effects. Providers also monitor patients' nonverbal behavior and reported affect, offering feedback to enhance engagement and perceived treatment quality.

Participants undergo MRI scanning, physiological monitoring, and behavioral assessments during Experiment 2. Multimodal physiological data-including ECG, respiration, skin conductance, photoplethysmography (PPG), and trans-radial electrical bioimpedance velocimetry (TRVE)-are collected using the BIOPAC 160 system.

ELIGIBILITY:
Inclusion Criteria:

'Doctors' are recruited from medical students at the Geisel School of Medicine and resident physicians at Dartmouth Hitchcock Medical Center (DHMC).

Exclusion Criteria:

* No self-reported current or history of depression, bipolar disorder, or other psychiatric diagnosis
* No self-reported current seizure disorder (i.e., seizure within past 10 years), or history of stroke or other major neurological diagnosis that can cause cognitive impairment
* No self-reported current chronic pain, or acute pain within three months of the study period
* No current migraine disorder (i.e., 15 headache days or more in 1 month)
* No use of central nervous system-effective medication or other medication for neurological/psychiatric treatment
* No self-reported substance abuse within the last six months
* No contraindication to MRI or tTIS (e.g., pregnancy, claustrophobia, pacemakers, ear/cochlear implants, shrapnel injuries, clips, or other ferromagnetic/electrical objects/devices, diagnosed brain abnormality such as tumor, or skin lesions on the scalp.)
* No contraindications for induced pain (e.g., no heart disease, high blood pressure, heart surgery, heart problems of any kind, severe asthma, respiratory problems of any kind, fibromyalgia, Raynaud's Syndrome or Disease, chronic pain, diabetes)
* Participants must be capable of performing experimental tasks (e.g., are able to read), are fluent or native speakers of English
* Participants must be able to tolerate the maximum level of thermal pain stimuli (for thermal stimuli)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 190 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2027-03-03 (Estimated)

PRIMARY OUTCOMES:
Cognitive effort ratings | 3-10 sec post-stimulus throughout testing sessions, with all sessions complete within 1 month
  Participants report cognitive effort after each trial on a Generalized Linear Magnitude scale (GLMS) with anchors of "No effort" and "Most effort imaginable". Raw units are on a 0-180 scale.
Subjective fear ratings | 3-10 sec post-stimulus throughout testing sessions, with all sessions complete within 1 month
  Participants report subjective fear experience after each trial on a well-validated Generalized Linear Magnitude scale (GLMS) with anchors of "No fear" and "Most intense fear imaginable". Raw units are on a 0-180 scale.
Pain ratings | 3-10 sec post-stimulus throughout testing sessions, with all sessions complete within 1 month
  Participants report subjective pain experience after each trial on a well-validated Generalized Linear Magnitude scale (GLMS) with anchors of "No pain" and "Most intense pain imaginable". Raw units are on a 0-180 scale.

SECONDARY OUTCOMES:
Electrodermal autonomic responses to painful heat, fear-related images and cognitive effort | Peri-stimulus throughout testing sessions, with all sessions complete within 1 month
  Skin conductance (EDA) is recorded continuously throughout test sessions and per-stimulus amplitude of canonical stimulus-locked EDA responses is reported in microsiemens (uS). Higher values indicate a higher EDA response.

CONTACTS AND LOCATIONS:
Locations (1):
- Dartmouth College, Department of Psychological and Brain Sciences, Hanover, New Hampshire, United States

REFERENCES:
- [Background] Acerbo E, Jegou A, Luff C, Dzialecka P, Botzanowski B, Missey F, Ngom I, Lagarde S, Bartolomei F, Cassara A, Neufeld E, Jirsa V, Carron R, Grossman N, Williamson A. Focal non-invasive deep-brain stimulation with temporal interference for the suppression of epileptic biomarkers. Front Neurosci. 2022 Aug 17;16:945221. doi: 10.3389/fnins.2022.945221. eCollection 2022. PMID 36061593
- [Background] Wessel MJ, Beanato E, Popa T, Windel F, Vassiliadis P, Menoud P, Beliaeva V, Violante IR, Abderrahmane H, Dzialecka P, Park CH, Maceira-Elvira P, Morishita T, Cassara AM, Steiner M, Grossman N, Neufeld E, Hummel FC. Noninvasive theta-burst stimulation of the human striatum enhances striatal activity and motor skill learning. Nat Neurosci. 2023 Nov;26(11):2005-2016. doi: 10.1038/s41593-023-01457-7. Epub 2023 Oct 19. PMID 37857774
- [Background] von Conta J, Kasten FH, Schellhorn K, Curcic-Blake B, Aleman A, Herrmann CS. Benchmarking the effects of transcranial temporal interference stimulation (tTIS) in humans. Cortex. 2022 Sep;154:299-310. doi: 10.1016/j.cortex.2022.05.017. Epub 2022 Jun 16. PMID 35839572
- [Background] Violante IR, Alania K, Cassara AM, Neufeld E, Acerbo E, Carron R, Williamson A, Kurtin DL, Rhodes E, Hampshire A, Kuster N, Boyden ES, Pascual-Leone A, Grossman N. Non-invasive temporal interference electrical stimulation of the human hippocampus. Nat Neurosci. 2023 Nov;26(11):1994-2004. doi: 10.1038/s41593-023-01456-8. Epub 2023 Oct 19. Erratum In: Nat Neurosci. 2023 Dec;26(12):2252. doi: 10.1038/s41593-023-01517-y. PMID 37857775
- [Background] Vassiliadis P, Beanato E, Popa T, Windel F, Morishita T, Neufeld E, Duque J, Derosiere G, Wessel MJ, Hummel FC. Non-invasive stimulation of the human striatum disrupts reinforcement learning of motor skills. Nat Hum Behav. 2024 Aug;8(8):1581-1598. doi: 10.1038/s41562-024-01901-z. Epub 2024 May 29. PMID 38811696
- [Background] Sandra DA, Olson JA, Langer EJ, Roy M. Presenting a sham treatment as personalised increases the placebo effect in a randomised controlled trial. Elife. 2023 Jul 5;12:e84691. doi: 10.7554/eLife.84691. PMID 37405829
- [Background] Grossman N, Bono D, Dedic N, Kodandaramaiah SB, Rudenko A, Suk HJ, Cassara AM, Neufeld E, Kuster N, Tsai LH, Pascual-Leone A, Boyden ES. Noninvasive Deep Brain Stimulation via Temporally Interfering Electric Fields. Cell. 2017 Jun 1;169(6):1029-1041.e16. doi: 10.1016/j.cell.2017.05.024. PMID 28575667